CLINICAL TRIAL: NCT00931723
Title: An International, Multicenter, Double-blind, Randomized, Placebo-controlled, Phase IV Study of the Safety and Efficacy of Lithium Versus Placebo as an Add on to SEROQUEL XR (Quetiapine Fumarate) in Adult Patients With Acute Mania
Brief Title: Adult Bipolar Mania
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D144AC00003
Record Dates: First submitted 2009-06-29; First posted 2009-07-02 (Estimated); Results first posted 2012-04-19 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-03

CONDITIONS: Acute Mania
Keywords: Acute Mania; Mania, Adults; Seroquel; Acute Mania in Adult Patients
MeSH Terms: conditions — Mania | interventions — Lithium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Seroquel XR and Lithium
  Interventions: Drug: Quetiapine fumarate XR; Drug: Lithium
- 2 (Placebo Comparator): Seroquel XR and placebo
  Interventions: Drug: Quetiapine fumarate XR; Drug: Placebo

INTERVENTIONS:
Drug: Quetiapine fumarate XR — Oral treatment, once daily, Day 1 = 300 mg, Day 2 and thereafter 600 mg. Dose might be adjusted as from Day 3 by the discretion of the investigator.
  Other Names: Seroquel XR
Drug: Lithium — Oral treatment, twice daily, Days 1 and 2 = 600 mg/day, Days 3-8 = 900 mg/day. Dose adjustment from day 9 to end of study will be at the discretion of the investigator.
  Arms: 1
Drug: Placebo — Oral treatment twice daily.
  Arms: 2

SUMMARY:
The purpose of this study is to determine if lithium 600-1800 mg/day is effective when added to quetiapine fumarate extended release (quetiapine XR or SEROQUEL® XR) 400-800 mg/day in treating acute mania and if so, how it compares with placebo (a non-active capsule, like a sugar pill, that looks like lithium).

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent before any study procedures are performed.
* The patient must have a documented clinical diagnosis for bipolar I disorder, including recent episode manic or mixed, and being male of females age 18-65 years, inclusive.
* Patients may be outpatients or inpatients at enrollment visit, but all patients must be inpatients when randomized and remain inpatients until discharged at the discretion of the investigator.

Exclusion Criteria:

* The patient can not have had up to 8 mood episodes during the past 12 months and not been continuously hospitalized for acute bipolar for up to 3 weeks immediately before participating in the study.
* The patient can not have a past diagnosis of stroke or medically documented transient ischemic attacks (TIA) or a history of seizure disorder, except for febrile convulsions.
* The patient must not have received electroconvulsive treatment (ECT) within 90 days before participating in the study and in the doctors judgement pose a current suicidal or homicidal risk.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2009-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Castiglione, Study Director — AstraZeneca; Michel Bourin, Professeur, Principal Investigator — Neurobiologie de l'anxiété et de la dépression Faculté de Médecine
Locations (65):
- Belgium (5):
  - Research Site, Montignies-sur-Sambre, Belgium
  - Research Site, Overpelt, Belgium
  - Research Site, Cedex, Cedex
  - Research Site, Dendermonde
  - Research Site, Tournai
- Bulgaria (7):
  - Research Site, Burgas, Bulgaria
  - Research Site, Radnevo, Bulgaria
  - Research Site, Cedex, Cedex
  - Research Site, Kazanlak
  - Research Site, Pazardzhik
  - Research Site, Plovdiv
  - Research Site, Sofia
- Germany (7):
  - Research Site, Cedex, Cedex
  - Research Site, Cologne, North Rhine-Westphalia
  - Research Site, Berlin, State of Berlin
  - Research Site, Berlin
  - Research Site, Mannheim
  - Research Site, München
  - Research Site, Nuremberg
- India (9):
  - Research Site, Visakhapatnam, Andh Prad
  - Research Site, Cedex, Cedex
  - Research Site, Ahmedabad, Gujarat
  - Research Site, Bangalore, Karna
  - Research Site, Mangalore, Karna
  - Research Site, Manipal, Karna
  - Research Site, Nashik, Mahara
  - Research Site, Jaipur, Rajasthan
  - Research Site, Kanpur, Uttar Prad
- Israel (6):
  - Research Site, Cedex, Cedex
  - Research Site, Bat Yam
  - Research Site, Beer Ya'acov
  - Research Site, Haifa
  - Research Site, Petah Tikva
  - Research Site, Tel Litwinsky
- Poland (8):
  - Research Site, Cedex, Cedex
  - Research Site, Bydgoszcz, Poland
  - Research Site, Choroszcz, Poland
  - Research Site, Gorlice
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lublin
  - Research Site, Poznan
- Russia (8):
  - Research Site, Cedex, Cedex
  - Research Site, Arkhangelsk
  - Research Site, Chita
  - Research Site, Kazan'
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Saratov
  - Research Site, Voronezh
- South Africa (7):
  - Research Site, Cedex, Cedex
  - Research Site, Bloemfontein, Free State
  - Research Site, Vereeniging, Free State
  - Research Site, Worcester, W Cape
  - Research Site, Cape Town
  - Research Site, Johannesburg
  - Research Site, Port Elizabeth
- Ukraine (8):
  - Research Site, Cedex, Cedex
  - Research Site, Kharkiv, Ukraine
  - Research Site, Kiev, Ukraine
  - Research Site, Dnipropetrovsk
  - Research Site, Donetsk
  - Research Site, Kiev
  - Research Site, Odesa
  - Research Site, Vinnitsia

REFERENCES:
- [Derived] Bourin MS, Severus E, Schronen JP, Gass P, Szamosi J, Eriksson H, Chandrashekar H. Lithium as add-on to quetiapine XR in adult patients with acute mania: a 6-week, multicenter, double-blind, randomized, placebo-controlled study. Int J Bipolar Disord. 2014 Nov 8;2:14. doi: 10.1186/s40345-014-0014-9. eCollection 2014. PMID 25505693

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter study was conducted between 24 June 2009 and 22 November 2010.
Pre-assignment Details: The study had an up to 28-day enrollment period (including a washout period lasting 7 to 28 days) and a 6-week double-blind treatment period. Patients were randomized to receive lithium 600 to 1800 mg/day+quetiapine XR 400 to 800 mg/day or placebo+quetiapine XR 400 to 800 mg/day.
Groups:
- Lithium+Quetiapine XR: Lithium 600 to 1800 mg/day+quetiapine XR 400 to 800 mg/day
- Placebo+Quetiapine XR: Placebo+quetiapine XR 400 to 800 mg/day
Period: Overall Study
Arm/Group | Lithium+Quetiapine XR | Placebo+Quetiapine XR
Started | 173 | 183
Completed | 147 | 144
Not Completed | 26 | 39
Not completed — Withdrawal by Subject | 11 | 13
Not completed — Adverse Event | 6 | 13
Not completed — Lithium found in blood | 0 | 1
Not completed — Condition under investigation worsened | 1 | 2
Not completed — Lost to Follow-up | 1 | 2
Not completed — Study-specific discontinuation criteria | 1 | 1
Not completed — Severe non-compliance to protocol | 2 | 0
Not completed — Safety reasons | 0 | 1
Not completed — Took prohibited concomitant medication | 0 | 1
Not completed — Lack or insufficient theraputic response | 2 | 5
Not completed — Sponsor decision | 1 | 0
Not completed — Late hospital discharge | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lithium+Quetiapine XR | Placebo+Quetiapine XR | Total
Number analyzed (Participants) | 173 | 183 | 356
Age Continuous [Mean (Standard Deviation); unit: Years] | 37.9 (12.71) | 38.8 (12.09) | 38.3 (12.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 62 | 134
  Male | 101 | 121 | 222

OUTCOME MEASURES:

1. Primary Outcome: Change in the Young Mania Rating Scale (YMRS) Total Score From Baseline to Final Assessment (Day 43)
Description: The YMRS total score ranges from 0 to 60 where higher scores indicate more severe mania, thus, a negative change (or decrease) from baseline indicates a reduction (or improvement) in manic symptoms. Total score ≤12 indicates remission (13-19=minimal symptoms; 20-25=mild mania, 26-37=moderate mania, 38-60=severe mania).
Time Frame: Change in YMRS total score from baseline to Day 43.
Population: 173/176 is modified intent to treat analysis set. The reason why is different from 173/183 is that there is 7 patients excluded from the analysis (1 patient who did not take study drug and 6 patients who did not have post treatment YMRS scores).
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Lithium+Quetiapine XR | Placebo+Quetiapine XR
Number analyzed (Participants) | 173 | 176
Scores on a scale | -22.8 (0.706) [lower limit 0.706] | -20.1 (0.711) [lower limit 0.711]

2. Secondary Outcome: The Number of Patients With Clinically Significant Response.
Description: The number of patients with clinically significant response (defined as ≥50% reduction from baseline to Day 43 in the YMRS total score) was calculated. The YMRS total score ranges from 0 to 60 where higher scores indicate more severe mania, thus, a negative change (or 50% reduction) from baseline indicates a reduction (or improvement) in manic symptoms.
Time Frame: 43 days (from baseline to Day 43)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Lithium+Quetiapine XR | Placebo+Quetiapine XR
Number analyzed (Participants) | 173 | 176
Participants | 137 | 120

3. Secondary Outcome: Remission
Description: The number of patients with clinically significant remission (defined as YMRS total score ≤12) from Days 8 to 43) was calculated.
  The Young Mania Rating Scale total score ranges from 0 to 60 where higher scores indicate more severe mania, thus, a negative change (or 50% reduction) from baseline indicates a reduction (or improvement) in manic symptoms. Total score ≤12 indicates remission (13-19=minimal symptoms; 20-25=mild mania, 26-37=moderate mania, 38-60=severe mania).
Time Frame: Days 8 to 43
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Lithium+Quetiapine XR | Placebo+Quetiapine XR
Number analyzed (Participants) | 173 | 176
Participants | 125 | 105

4. Secondary Outcome: Change From Baseline to Day 43 in CGI-BP-S (Clinical Global Impressions for Bipolar Disorder-Severity of Illness)
Description: The CGI-BP-S scale rates the severity of the patient's illness at the time of assessment and is scored from 1 to 7 (1=normal, not ill to 7=very severely ill). Higher CGI-BP-S scores indicate greater illness severity.
Time Frame: Change from baseline to Day 43.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Lithium+Quetiapine XR | Placebo+Quetiapine XR
Number analyzed (Participants) | 173 | 176
Scores on a scale | -2.5 (0.079) [lower limit 0.079] | -2.2 (0.080) [lower limit 0.080]

5. Secondary Outcome: Change From Baseline to Day 43 in CGI-BP-C (Clinical Global Impressions for Bipolar Disorder-Change From Preceding Phase)
Description: The CGI-BP-C scale rates how much the patient's illness has improved or worsened compared to the phase immediately preceding treatment and is scored on a scale from 1 to 8 (1=very much improved to 7=very much worse; 8=not applicable). A missing score will be used when a scale scored as 8 (not applicable). CGI-BP-C scores >4 indicate worsening, while scores <4 indicate improvement.
Time Frame: Change from baseline to Day 43
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Lithium+Quetiapine XR | Placebo+Quetiapine XR
Number analyzed (Participants) | 173 | 176
Scores on a scale | 1.7 (0.085) [lower limit 0.085] | 1.9 (0.086) [lower limit 0.086]

6. Secondary Outcome: Improvement of Overall Bipolar Illness
Description: The number of patients with a CGI-BP-C of "Much" or "Very much" improved in overall bipolar illness assessment at Day 43 was calculated.
  The CGI-BP-C scale rates how much the patient's illness has improved or worsened compared to the phase immediately preceding treatment and is scored on a scale from 1 to 8 (1=very much improved to 7=very much worse; 8=not applicable). A missing score will be used when a scale scored as 8 (not applicable). CGI-BP-C scores >4 indicate worsening, while scores <4 indicate improvement.
Time Frame: Day 43.
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Lithium+Quetiapine XR | Placebo+Quetiapine XR
Number analyzed (Participants) | 173 | 176
Participants | 134 | 125

7. Secondary Outcome: Change From Baseline to Day 43 in Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score
Description: The MADRS is a 10-item scale that evaluates depressive symptoms. Each MADRS item is rated on a 0 to 6 scale. Higher MADRS scores indicate higher levels of depressive symptoms.
Time Frame: Change from baseline to Day 43.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Lithium+Quetiapine XR | Placebo+Quetiapine XR
Number analyzed (Participants) | 173 | 176
Scores on a scale | -4.8 (0.366) [lower limit 0.366] | -4.1 (0.368) [lower limit 0.368]

8. Secondary Outcome: Change From Baseline to Day 43 in Positive and Negative Syndrome Scale (PANSS) Total Score
Description: The PANSS is a 30-item scale designed to assess various symptoms of schizophrenia and are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS total score is the sum of all 30 individual-item scores and ranges from 30 to 210.A negative change (or decrease) from baseline indicates a reduction (or improvement) in symptoms.
Time Frame: Change from baseline to Day 43
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Lithium+Quetiapine XR | Placebo+Quetiapine XR
Number analyzed (Participants) | 173 | 176
Scores on a scale | -19.2 (0.914) [lower limit 0.914] | -15.6 (0.914) [lower limit 0.914]

9. Secondary Outcome: Change From Baseline to Day 43 in PANSS Activation Subscale Score
Description: The PANSS is a 30-item scale designed to assess various symptoms of schizophrenia and are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS activation subscale score for effect on agitation and aggression is the sum of 6 PANSS individual items (ie, hostility, poor impulse control, excitement, uncooperativeness, poor rapport and tension) and ranges from 6 to 42. A negative change (or decrease) from baseline indicates a reduction (or improvement) in symptoms.
Time Frame: Change from baseline to Day 43
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Lithium+Quetiapine XR | Placebo+Quetiapine XR
Number analyzed (Participants) | 173 | 176
Scores on a scale | -7.1 (0.281) [lower limit 0.281] | -5.9 (0.283) [lower limit 0.283]

10. Secondary Outcome: Change From Baseline to Day 43 in PANSS Positive Subscale Score
Description: The PANSS is a 30-item scale designed to assess various symptoms of schizophrenia and are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS positive subscale score is the sum of the 7 positive item scores (ie, delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution and hostility) and ranges from 7 to 49. A negative change (or decrease) from baseline indicates a reduction (or improvement) in symptoms.
Time Frame: Change from baseline to Day 43
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Lithium+Quetiapine XR | Placebo+Quetiapine XR
Number analyzed (Participants) | 173 | 176
Scores on a scale | -8.1 (0.316) [lower limit 0.316] | -7.0 (0.316) [lower limit 0.316]

11. Secondary Outcome: Change From Baseline to Day 43 in Each YMRS Item Score No. 1
Description: The YMRS assesses severity of mania in bipolar disorder. It rates 4 core items from 0 to 8 (0=normal); the other 7 items are rated from 0 to 4 (0=normal). This analysis is for Item 1 (Elevated mood) which ranges from 0 to 4 where higher scores indicate more severe symptoms, thus, a negative change (or decrease) from baseline indicates a reduction (or improvement) in symptoms.
Time Frame: Change from baseline to Day 43
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Lithium+Quetiapine XR | Placebo+Quetiapine XR
Number analyzed (Participants) | 173 | 176
Scores on a scale | -1.8 (0.079) [lower limit 0.079] | -1.6 (0.080) [lower limit 0.080]

12. Secondary Outcome: Change From Baseline to Day 43 in Each YMRS Item Score No. 2
Description: The YMRS assesses severity of mania in bipolar disorder. It rates 4 core items from 0 to 8 (0=normal); the other 7 items are rated from 0 to 4 (0=normal). This analysis is for Item 2 (increased motor activity-energy) which ranges from 0 to 4 where higher scores indicate more severe symptoms, thus, a negative change (or decrease) from baseline indicates a reduction (or improvement) in symptoms.
Time Frame: Change from baseline to Day 43
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Lithium+Quetiapine XR | Placebo+Quetiapine XR
Number analyzed (Participants) | 173 | 176
Scores on a scale | -1.9 (0.071) [lower limit 0.071] | -1.7 (0.072) [lower limit 0.072]

13. Secondary Outcome: Change From Baseline to Day 43 in Each YMRS Item Score No. 3
Description: The YMRS assesses severity of mania in bipolar disorder. It rates 4 core items from 0 to 8 (0=normal); the other 7 items are rated from 0 to 4 (0=normal). This analysis is for Item 3 (sexual interest) which ranges from 0 to 4 where higher scores indicate more severe symptoms, thus, a negative change (or decrease) from baseline indicates a reduction (or improvement) in symptoms.
Time Frame: Change from baseline to Day 43
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Lithium+Quetiapine XR | Placebo+Quetiapine XR
Number analyzed (Participants) | 173 | 176
Scores on a scale | -1.3 (0.063) [lower limit 0.063] | -1.1 (0.064) [lower limit 0.064]

14. Secondary Outcome: Change From Baseline to Day 43 in Each YMRS Item Score No. 4
Description: The YMRS assesses severity of mania in bipolar disorder. It rates 4 core items from 0 to 8 (0=normal); the other 7 items are rated from 0 to 4 (0=normal). This analysis is for Item 4 (sleep) which ranges from 0 to 4 where higher scores indicate more severe symptoms, thus, a negative change (or decrease) from baseline indicates a reduction (or improvement) in symptoms.
Time Frame: Change from baseline to Day 43
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Lithium+Quetiapine XR | Placebo+Quetiapine XR
Number analyzed (Participants) | 173 | 176
Scores on a scale | -2.0 (0.085) [lower limit 0.085] | -1.8 (0.086) [lower limit 0.086]

15. Secondary Outcome: Change From Baseline to Day 43 in Each YMRS Item Score No. 5
Description: The YMRS assesses severity of mania in bipolar disorder. It rates 4 core items from 0 to 8 (0=normal); the other 7 items are rated from 0 to 4 (0=normal). This analysis is for Item 5 (Irritability) which ranges from 0 to 8 where higher scores indicate more severe symptoms, thus, a negative change (or decrease) from baseline indicates a reduction (or improvement) in symptoms.
Time Frame: Change from baseline to Day 43
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Lithium+Quetiapine XR | Placebo+Quetiapine XR
Number analyzed (Participants) | 173 | 176
Scores on a scale | -3.1 (0.109) [lower limit 0.109] | -2.8 (0.110) [lower limit 0.110]

16. Secondary Outcome: Change From Baseline to Day 43 in Each YMRS Item Score No. 6
Description: The YMRS assesses severity of mania in bipolar disorder. It rates 4 core items from 0 to 8 (0=normal); the other 7 items are rated from 0 to 4 (0=normal). This analysis is for Item 6 (speech-rate and amount) which ranges from 0 to 8 where higher scores indicate more severe symptoms, thus, a negative change (or decrease) from baseline indicates a reduction (or improvement) in symptoms.
Time Frame: Change from baseline to Day 43
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Lithium+Quetiapine XR | Placebo+Quetiapine XR
Number analyzed (Participants) | 173 | 176
Scores on a scale | -3.1 (0.116) [lower limit 0.116] | -2.9 (0.118) [lower limit 0.118]

17. Secondary Outcome: Change From Baseline to Day 43 in Each YMRS Item Score No. 7
Description: The YMRS assesses severity of mania in bipolar disorder. It rates 4 core items from 0 to 8 (0=normal); the other 7 items are rated from 0 to 4. This analysis is for Item 7 (language-thought disorder) which ranges from 0 to 4 where higher scores indicate more severe symptoms, thus, a negative change (or decrease) from baseline indicates a reduction (or improvement) in symptoms.
Time Frame: Change from baseline to Day 43
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Lithium+Quetiapine XR | Placebo+Quetiapine XR
Number analyzed (Participants) | 173 | 176
Scores on a scale | -1.5 (0.071) [lower limit 0.071] | -1.4 (0.072) [lower limit 0.072]

18. Secondary Outcome: Change From Baseline to Day 43 in Each YMRS Item Score No. 8
Description: The YMRS assesses severity of mania in bipolar disorder. It rates 4 core items from 0 to 8 (0=normal); the other 7 items are rated from 0 to 4. This analysis is for Item 8 (content) which ranges from 0 to 8 where higher scores indicate more severe symptoms, thus, a negative change (or decrease) from baseline indicates a reduction (or improvement) in symptoms.
Time Frame: Change from baseline to Day 43
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Lithium+Quetiapine XR | Placebo+Quetiapine XR
Number analyzed (Participants) | 173 | 176
Scores on a scale | -3.1 (0.132) [lower limit 0.132] | -2.9 (0.133) [lower limit 0.133]

19. Secondary Outcome: Change From Baseline to Day 43 in Each YMRS Item Score No. 9
Description: The YMRS assesses severity of mania in bipolar disorder. It rates 4 core items from 0 to 8 (0=normal); the other 7 items are rated from 0 to 4. . This analysis is for Item 9 (disruptive-aggressive behavior) which ranges from 0 to 8 where higher scores indicate more severe symptoms, thus, a negative change (or decrease) from baseline indicates a reduction (or improvement) in symptoms.
Time Frame: Change from baseline to Day 43
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Lithium+Quetiapine XR | Placebo+Quetiapine XR
Number analyzed (Participants) | 173 | 176
Scores on a scale | -2.5 (0.088) [lower limit 0.088] | -2.1 (0.089) [lower limit 0.089]

20. Secondary Outcome: Change From Baseline to Day 43 in Each YMRS Item Score No. 10
Description: The YMRS assesses severity of mania in bipolar disorder. It rates 4 core items from 0 to 8 (0=normal); the other 7 items are rated from 0 to 4. This analysis is for Item 10 (appearance) which ranges from 0 to 4 where higher scores indicate more severe symptoms, thus, a negative change (or decrease) from baseline indicates a reduction (or improvement) in symptoms.
Time Frame: Change from baseline to Day 43
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Lithium+Quetiapine XR | Placebo+Quetiapine XR
Number analyzed (Participants) | 173 | 176
Scores on a scale | -1.1 (0.057) [lower limit 0.057] | -1.0 (0.057) [lower limit 0.057]

21. Secondary Outcome: Change From Baseline to Day 43 in Each YMRS Item Score No. 11
Description: The YMRS assesses severity of mania in bipolar disorder. It rates 4 core items from 0 to 8 (0=normal); the other 7 items are rated from 0 to 4. This analysis is for Item 11 (insight) which ranges from 0 to 4 where higher scores indicate more severe symptoms, thus, a negative change (or decrease) from baseline indicates a reduction (or improvement) in symptoms.
Time Frame: Change from baseline to Day 43
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Lithium+Quetiapine XR | Placebo+Quetiapine XR
Number analyzed (Participants) | 173 | 176
Scores on a scale | -1.4 (0.069) [lower limit 0.069] | -1.2 (0.070) [lower limit 0.070]

ADVERSE EVENTS:
Arm/Group | Lithium+Quetiapine XR | Placebo+Quetiapine XR
Serious Adverse Events (participants affected / at risk) | 4/173 | 8/183
Other Adverse Events (participants affected / at risk) | 106/173 | 83/183
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lithium+Quetiapine XR (N=173) | Placebo+Quetiapine XR (N=183)
Mania (Psychiatric disorders) | 3 | 6
Aggression; Hostility (Psychiatric disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
No Therapeutic Response (Investigations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lithium+Quetiapine XR (N=173) | Placebo+Quetiapine XR (N=183)
Tremor (Nervous system disorders) | 27 | 9
Somnolence (Nervous system disorders) | 22 | 10
Dizziness (Nervous system disorders) | 11 | 8
Headache (Nervous system disorders) | 9 | 11
Sedation (Nervous system disorders) | 5 | 3
Dysarthria (Nervous system disorders) | 4 | 2
Constipation (Gastrointestinal disorders) | 16 | 16
Dry Mouth (Gastrointestinal disorders) | 14 | 14
Diarrhoea (Gastrointestinal disorders) | 8 | 2
Vomiting (Gastrointestinal disorders) | 8 | 0
Nausea (Gastrointestinal disorders) | 5 | 3
Insomnia (Psychiatric disorders) | 11 | 12
Pyrexia (General disorders) | 10 | 9
Weight Increased (Investigations) | 2 | 5
Increased Appetite (Metabolism and nutrition disorders) | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other